CLINICAL TRIAL: NCT01785004
Title: Interrelationship of Vitamin D Supplementation, Adiposity and CVD Risk Factors in a Randomized Clinical Trial
Brief Title: Vitamin D and Omega-3 Adiposity Trial (VITAL Adiposity)
Acronym: VITAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Jacqueline Suk Danik, MD, DrPH, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2012P001304; 12GRNT11980009 (Other Grant/Funding Number: AHA)
Record Dates: First submitted 2013-01-23; First posted 2013-02-06 (Estimated); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Adiposity
Keywords: Adiposity; Body composition; Vitamin D; Adipokines; Omega-3 fatty acid
MeSH Terms: conditions — Obesity | interventions — Cholecalciferol; Fatty Acids, Omega-3; Fish Oils; Omacor; Eicosapentaenoic Acid; Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Vitamin D + fish oil (Active Comparator): Vitamin D3 (cholecalciferol), 2000 IU per day and 840 mg of marine omega-3 fatty acids (465 mg of eicosapentaenoic acid [EPA] and 375 mg of docosahexaenoic acid [DHA])
  Interventions: Dietary Supplement: Vitamin D3 (cholecalciferol), 2000 IU per day; Drug: omega-3 fatty acids (fish oil)
- Vitamin D + fish oil placebo (Active Comparator): Vitamin D3 (cholecalciferol), 2000 IU per day and fish oil placebo
  Interventions: Dietary Supplement: Vitamin D3 (cholecalciferol), 2000 IU per day
- Vitamin D placebo + fish oil (Active Comparator): Vitamin D placebo and 840 mg of marine omega-3 fatty acids (465 mg of eicosapentaenoic acid [EPA] and 375 mg of docosahexaenoic acid [DHA])
  Interventions: Drug: omega-3 fatty acids (fish oil)
- Vitamin D placebo + fish oil placebo (Placebo Comparator): Vitamin D placebo and fish oil placebo
  Interventions: Dietary Supplement: Vitamin D3 (cholecalciferol), 2000 IU per day; Drug: omega-3 fatty acids (fish oil)

INTERVENTIONS:
Dietary Supplement: Vitamin D3 (cholecalciferol), 2000 IU per day — cholecalciferol
  Arms: Vitamin D + fish oil; Vitamin D + fish oil placebo; Vitamin D placebo + fish oil placebo
Drug: omega-3 fatty acids (fish oil)
  Other Names: Omacor, 1 capsule a day.; Each capsure of Omacor contains 840 milligrams of marine omega-3 fatty acid; (465 mg of eicosapentaenoic acid [EPA] and 375 mg of docosahexaenoic acid [DHA]).
  Arms: Vitamin D + fish oil; Vitamin D placebo + fish oil; Vitamin D placebo + fish oil placebo

SUMMARY:
The VITamin D and OmegA-3 TriaL (VITAL; NCT 01169259) is a randomized clinical trial in 20,000 U.S. men and women investigating whether taking daily dietary supplements of vitamin D3 (2000 IU) or omega-3 fatty acids (1 gram of omega-3 fatty acids) reduces the risk of developing cancer, heart disease, and stroke in people who do not have a prior history of these illnesses. This ancillary study (VITAL Adiposity) is being conducted among participants in VITAL and will examine the effect of vitamin D or fish oil on changes in body composition and adiposity (baseline compared to 2 year, as measured by anthropometric indices, total and regional body fat and adipokines) and assess whether changes in cardiovascular risk factors (lipids, glucose tolerance, blood pressure) are mediated by these parameters. How achieved 25(OH)D levels are affected by body composition and body mass will also be assessed.

DETAILED DESCRIPTION:
Observational studies suggest that low 25-hydroxyvitamin D (25(OH)D) levels are associated with high BMI and fat mass (FM), but it is unknown whether vitamin D supplementation can alter body composition or adiposity. Despite enthusiasm for the use of vitamin D supplements to reduce FM, the hypothesis that vitamin D can modify adiposity remains unproven. Finding strategies to prevent obesity is of critical public health importance due to the high prevalence of overweight/obesity and its role in causing diabetes, hypertension, dyslipidemia, cardiovascular disease (CVD), among others. Observational studies also link low 25(OH)D levels to CVD risk factors related to obesity, but sequestration of vitamin D in fat tissue may be a confounding factor. The effects of vitamin D supplementation on body composition, adiposity and CVD risk factors are best tested in a randomized clinical trial (RCT), and according to the Institute of Medicine (IOM) 2011 report, more data from randomized clinical trials on these outcomes are needed. Previous trials of vitamin D have been limited by the inability to separate effects of supplemental calcium from vitamin D, small sample size, insufficient vitamin D dose, failure to monitor 25(OH)D levels or inadequate ascertainment of body composition. The NIH-funded VITamin D and OmegA-3 TriaL (VITAL) (1 U01 CA138962) affords a unique and cost-effective opportunity to investigate the effect of vitamin D on changes in body composition and to assess whether changes in CVD risk factors are mediated, at least in part, by these parameters. VITAL is a large-scale, randomized, primary prevention trial testing 2000 IU/d vitamin D3 (cholecalciferol) and 1 g/day omega-3 fatty acids (840 mg EPA+DHA in 1.3:1 ratio) in a 2x2 factorial design among 20,000 men and women (≥50 and ≥55 years, respectively), with mean participant follow-up of 5 years for CVD and cancer. This ancillary study will address understudied areas and two overarching hypotheses that vitamin D supplementation (1) lowers total and regional (trunkal and abdominal/androidal) body fat as measured by dual x-ray absorptiometry (DXA) scans, improving biomarkers of adiposity (leptin, adiponectin) and (2) impacts CVD risk factors, at least in part through adiposity. The investigators also seek to define how circulating achieved 25(OH)D levels, due to supplementation, may be affected by body composition and BMI, thus elucidating how adiposity, BMI, and body composition (total and regional) may influence vitamin D intake needs in the population. To critically evaluate these hypotheses, the investigators will examine a representative, randomized subcohort of 1000 racially diverse VITAL participants (25% African American) over two years.

ELIGIBILITY:
Inclusion criteria:

* Participants in VITAL (NCT 01169259) who are willing to participate in this ancillary study and undergo DXA evaluation (baseline and 2 years)

Exclusion criteria:

* Inability to travel to the Clinical and Translational Science Center in Boston where imaging, anthropometric measurements, and blood work will be performed.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2012-07; Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Body Composition | 2 years
  We will measure by DXA, changes in body composition (i) total body fat and lean mass, (ii) regional and standardized body fat and lean mass (trunkal, androidal (abdominal), appendicular (limb) and derived ratios (trunk/limb; android/gynoid)) among those randomized to vitamin D supplementation vs. those randomized to placebo.

SECONDARY OUTCOMES:
Anthropometric Measurements | 2 years
  We will perform and compare changes in anthropometric measurements, including BMI, waist circumference and waist-hip ratio.
Mediation of CVD risk factors by body composition | 2 years
  We will compare 2 year changes in CVD risk factors: (lipids [triglycerides, HDL, LDL]), glucose homeostasis (hemoglobin A1c, glucose, insulin, HOMA-IR) and blood pressure between treatment groups, and assess whether changes in body composition mediate any treatment effects.
Adipokines | 2 years
  Among 200 participants, we will assess effect of vitamin D supplementation on adipokines to assess for 2-year changes among those randomized to supplementation vs. placebo.
Achieved 25(OH)D level | 2 years
  We will assess whether achieved 25(OH)D levels with supplementation are affected by baseline and change in body composition and BMI.

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline S. Danik, MD, DrPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- See also: Related Info — http://www.vitalstudy.org/